CLINICAL TRIAL: NCT05367544
Title: Equity in Prevention and Progression of Hypertension by Addressing Barriers to Nutrition and Physical activitY
Acronym: EPIPHANY
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Andrea Cherrington, MD, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-300009015
Record Dates: First submitted 2022-04-12; First posted 2022-05-10 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Prehypertension; Hypertension; Blood Pressure
MeSH Terms: conditions — Prehypertension; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health Education & Peer Coaching (Experimental): Participants will have access to online health education materials and will also be matched with a community health worker who will offer support through peer coaching
  Interventions: Behavioral: Health Education; Behavioral: Individual-Level Peer Support; Behavioral: Community-Level Peer Support
- Health Education Only (Active Comparator): Participants will have access to online health education materials but will not receive individualized peer support
  Interventions: Behavioral: Health Education; Behavioral: Community-Level Peer Support

INTERVENTIONS:
Behavioral: Health Education — All participants will receive education regardless of randomization status. On the day of enrollment, participants will be invited to attend education modules focused on HTN risk, diet, physical activity, stress management, and goal setting. Participants will also have access to culturally relevant, weekly online sessions, alternating between cooking shows and exercise
Behavioral: Individual-Level Peer Support — Participants will receive bi-weekly peer support calls for 6 months, followed by monthly calls for another 6 months.
  Arms: Health Education & Peer Coaching
Behavioral: Community-Level Peer Support — Church Leadership in churches randomized to intervention will identify 2-3 Peer Health Advocates from the church who will receive training on ways to promote a culture of health, encouraging church members to attend on-line cooking shows and exercise sessions. After training, these individuals will also work with Church Leadership to form a committee that will develop a project (e.g., community food pantry, farmer's market, Zumba instruction, small church gym) aimed at overcoming structural barriers to healthy behaviors. Each church will receive a small stipend for their project. Churches randomized to education alone will receive the community-level intervention after 12 months of participation in the study (delayed intervention)

SUMMARY:
The goal of this study is to test an intervention to prevent high blood pressure among rural, Black adults living in Alabama. Black adults in this region have one of the highest rates of high blood pressure in the US. Eating fruits and vegetables and exercising daily lowers the chance of getting high blood pressure. Many problems get in the way of eating a healthy diet and exercising like a lack of grocery stores with fresh foods, few gyms, little money, lack of transportation, and limited support for keeping healthy habits. One place where many Black adults in rural Alabama meet weekly and feel supported is their church. The investigators will connect with 30 churches in rural Alabama. The investigators plan to hold health fairs to find 12 Black adults from each church with blood pressure that is higher than normal but not high enough to need blood pressure lowering medications. The investigators will randomly select 15 churches to get group health education and tablets to access online cooking shows and exercise classes. Adults in the other 15 churches will get support from a health coach over the telephone to help set and meet diet and physical activity goals as well as the group health education and tablets to access online cooking shows and exercise classes. In this study, the investigators will ask church members to sign up to be a health coach. These 15 churches will also get money to help bring healthy foods and/or physical activity opportunities to their communities. The investigative team will train 2 to 3 of their church members to learn how to coach others to eat more healthy food and be more physically active. This study answers two questions. 1) Will this intervention designed to reduce barriers to a healthy lifestyle lower blood pressure among rural, Black adults? 2) Can churches and participants complete the whole two-year study, and can the intervention be used in other communities in a cost-effective way to improve blood pressure? This project will add to the health equity mission of the American Heart Association by finding out if an intervention using health coaches lowers blood pressure among rural Black adults.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as Black/African American
* Mean systolic blood pressure 120-139mmHg OR diastolic blood pressure 80-89mmHg

Exclusion Criteria:

1. Mean systolic blood pressure greater than or equal to140 mm Hg, or mean diastolic blood pressure greater than or equal to 90 mm Hg
2. Currently taking antihypertensive medication
3. Self-reported history of hypertension outside of pregnancy
4. Known pregnancy
5. Self-reported history of cardiovascular disease
6. Age ≥65 years or self-reported history of chronic kidney disease, or diabetes, if systolic blood pressure ≥ 130 mm Hg or diastolic blood pressure ≥ 80
7. Planning to move out of the county within the next 18 months
8. Not having a cellular phone or landline
9. Inability to speak English

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 528 (Estimated)
Dates: Start 2022-08-13 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Incident Blood Pressure | Baseline, 6 months,12 months, 18 months
  Change in systolic blood pressure and diastolic blood pressure

SECONDARY OUTCOMES:
Fruit/Vegetable/Fiber Intake | Baseline, 6 months,12 months, 18 months
  Change in consumption of fruits, vegetables, and fiber rich foods
Physical Activity | Baseline, 6 months,12 months, 18 months
  Change in days per week participant participates in moderate and/or vigorous physical activity
Alcohol use | Baseline, 6 months,12 months, 18 months
  Change in consumption of alcoholic beverages
Smoking | Baseline, 6 months,12 months, 18 months
  Change in frequency in use of tobacco problems

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama At Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD with other researchers